CLINICAL TRIAL: NCT06291597
Title: VapALERT: A Prospective, Exploratory and Adaptive Cohort Study to Identify Symptomatic and Asymptomatic Pulmonary and Cardiovascular Effects of Vaping
Brief Title: Vaping Adverse Lung and Heart Events Cohort
Acronym: VapALERT
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Sponsor
Other Study IDs: 22071
Record Dates: First submitted 2023-10-07; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Vaping; Electronic Cigarette Use
Keywords: Vaping; Vape; Electronic cigarette; Electronic and vaping acute lung injury; EVALI
MeSH Terms: conditions — Vaping; Lung Injury | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat obtained from plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Daily electronic cigarette users: Participants must use their vaping device everyday at time of enrollment.
  Interventions: Other: Vaping

INTERVENTIONS:
Other: Vaping — Participants use their vaping products at their own discretion and their intake is monitored via questionnaires.

SUMMARY:
This prospective study assesses the pulmonary and cardiovascular effets of vaping in adult electronic cigarette users with biannual visits and a 5-year follow-up.

DETAILED DESCRIPTION:
Daily vaping device users will be recruited in the Quebec City metropolitan area. Subjects will be asked to perform pulmonary function tests (spirometry, oscillometry, plethysmography, methacholine provocation) every 6 months for a 5-year follow up. Subjects will also answer a questionnaire assessing their vaping, tobacco and cannabis smoking habits, as well as their perceived respiratory symptoms. Blood draws and sputum inductions will be performed for cell counts and to measure inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Daily electronic cigarette user
* No respiratory infection in the 4 weeks before a visit

Exclusion Criteria:

* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We seek to recruit 250 volunteers from the community with twice-a-year visits for a 5-year follow-up. We will recruit healthy volunteers as well as volunteers who have been previously diagnosed with chronic illness.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants who vape daily with impaired lung volumes. | Every 6 months for 5 years
  Participants will perform plethysmography assessments to measure changes in lung volumes. Data will be expressed as a percentage of predicted values.
Number of participants who vape daily with impaired lung diffusion capacity. | Every 6 months for 5 years
  Participants will perform diffusion capacity of the lung for carbon monoxide (DLCO) measures to assess changes in lung diffusion capacity. Data will be expressed as a percentage of predicted values.
Number of participants who vape daily with impaired spirometry. | Every 6 months for 5 years
  Participants will perform spirometry tests measures to assess changes in forced expiratory lung volumes. Data will be expressed as a percentage of predicted values.
Number of participants who vape daily with airway hyperresponsiveness. | Every 6 months for 5 years
  Participants will perform methacholine provocation challenge measures to assess changes in airway hyperresponsiveness. Data will be expressed as the methacholine concentration inducing a fall of 20% of forced expiratory volume in the first second assessed (PC20).
Number of participants who vape daily with changes in blood cell count. | Every 6 months for 5 years
  Participants will perform a blood draw to assess blood cell count. Data will be expressed as a percentage of eosinophils, neutrophils, macrophages and lymphocytes of the total cell count.
Number of participants who vape daily with changes in sputum cell count. | Every 6 months for 5 years
  Participants will perform sputum inductions to assess cell count in the sputum. Data will be expressed as a percentage of eosinophils, neutrophils, macrophages and lymphocytes of the total cell count.
Vaping, tobacco and cannabis smoking habits of participants. | Every 3 months for 5 years
  Participants will complete questionnaires assessing their vaping habits, tobacco smoking and cannabis smoking history.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu C Morissette, PhD, Principal Investigator — Laval University
Locations (1):
- IUCPQ-UL, Québec, Canada

IPD SHARING:
Plan to Share IPD: No